CLINICAL TRIAL: NCT00736541
Title: Investigation of the Efficacy of N-acetylcysteine (NAC) to Protect Against Hepato-renal Ischemia-reperfusion Injury in Patients Undergoing Orthotopic Liver Transplantation
Brief Title: N-acetylcysteine in Liver Transplantation
Acronym: NAC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ibtesam Hilmi (Other)
Responsible Party: Sponsor-Investigator, Ibtesam Hilmi, Professor, University of Pittsburgh
Organization: University of Pittsburgh (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: N-acetylcysteine in OLT
Record Dates: First submitted 2008-08-14; First posted 2008-08-18 (Estimated); Last update posted 2023-04-28 (Actual); Status verified 2023-04

CONDITIONS: End Stage Liver Failure
Keywords: ARF; OLT; NAC; I/R injury
MeSH Terms: interventions — Acetylcysteine; Glutathione; Cystatin C; prostaglandin R2 D-isomerase

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- 2 (Experimental)
  Interventions: Drug: N-acetylcysteine

INTERVENTIONS:
Drug: N-acetylcysteine — The patients in the NAC group will receive a loading dose of 140 mg/kg IV of NAC over one hour at the start of the surgery. Thereafter, NAC will be repeated every 4 hours at a dose of 70 mg/kg IV, for a total of 13 doses
  Other Names: NAC, GSH, cystatin-c, beta-trace

SUMMARY:
N-acetylcysteine (NAC) is used to treat Tylenol toxicity. NAC is a rich source of the sulfhydryl group (SH) which is important for replenishing the body's glutathione stores. Glutathione acts as a free radical scavenger, to decrease the damage that would be caused by those toxic radicals. Patients who undergo orthotopic liver transplantation (OLT) have a high incidence of post-operative renal dysfunction. The most common etiology of post-operative renal dysfunction is related to high levels of toxic free radicals. Free radicals may contribute to primary liver graft failure or delayed liver graft function.

Specific Aims & Objectives:

The primary objective of this study is to evaluate the efficacy of NAC in improving liver graft performance and lowering the incidence of post-operative renal dysfunction. The secondary objectives are to investigate the effect of NAC on endogenous glutathione body stores and its effect on FK506 induced toxicity.

DETAILED DESCRIPTION:
This is a randomized, double-blind placebo-controlled study that investigates the use of NAC during and after OLT. A total of 100 patients will be recruited. Fifty will receive a placebo (normal saline) and the other fifty will receive NAC. The patients in the NAC group will receive a loading dose of 140 mg/kg IV of NAC over one hour at the start of the surgery. Thereafter, NAC will be repeated every 4 hours at a dose of 70 mg/kg IV, for a total of 13 doses. The placebo group will receive an equal volume of a normal saline infusion for 13 doses. Both groups will be followed for one year after their OLT. The following data will be recorded and collected: liver function tests, renal function tests, liver graft survival rate, patient survival, serum level of glutathione (GSH-PX/GR), duration of hospital and ICU stay. To evaluate the accuracy of calculated serum creatinine clearance (CSCC) in predicating the renal performance in OLT patients, another two serum markers will be estimated. The 1st one is Cystatin-C and the 2nd is Beta-trace. The data from CSCC, cystatin-C and beta-trace will be compared to find out which is the best marker in between these three tests to predicate the renal function. The data will be recorded daily for the first week after the surgery, then on days 14, 21, 30, 90, 180 and finely at the end of the first year after the OLT. Statistical analysis of the data will be performed at the conclusion of the study period to determine the difference in the outcome and morbidity and mortality between the two groups.

Objective and Specific Aims

Objectives:

* Assess the efficacy of NAC to preserve liver graft function and to improve patient/graft survival following orthotopic liver transplantation.
* Assess the efficacy of NAC to preserve kidney function in the patients undergoing OLT.

Primary Aims:

* Severity of the post reperfusion syndrome (PRS) will be compared in both groups by assessing hemodynamic parameters and the need for vasopressor support in the neohepatic stage.
* Liver graft function, the incidence of primary non-function and delayed function in both the treatment and placebo groups, will be assessed with post-operative liver function tests (ALT, AST, serum bilirubin, PT/INR, APTT, lactate, etc). Liver function tests will be assessed at one month, three month, six month and at one year following the OLT.
* The duration of ICU and hospital stays will be compared between the two groups.
* Survival rate (patient/graft) between the treatment and placebo groups will be compared at 1 month, 3 months, 6 months and 1 year.
* Renal function will be compared in the treatment and placebo groups by assessing the following parameters during and after liver transplantation: urine output (ml/24 hours), serum creatinine and BUN, calculated creatinine clearance.
* The incidence of postoperative acute renal failure (ARF) and the extent and duration of renal dysfunction will be compared between the treatment and the placebo groups.

Secondary Aims:

* Investigating the effect of NAC on the endogenous glutathione peroxides/glutathione reductase (GSH-PX/GR) body stores in patients undergoing OLT.
* Investigating the effect of NAC on FK506 induced toxicity.
* Investigating the accuracy of two new markers for evaluating the renal function and glomerular filtration rate and compare them to CSCC.

ELIGIBILITY:
Inclusion Criteria:

* Male or female patients age of 18 years
* Patients undergoing cadaveric liver transplant for the first time
* Patients with normal serum creatinine < 1- 1.2 mg/dl or creatinine clearance 97-140 ml/min and patients with mild renal dysfunction with serum creatinine of (2-2.5 mg/dl) or creatinine clearance 85-125 ml/min
* All patients will sign informed consent

Exclusion Criteria:

* Allergy to NAC
* Patients with history of asthma
* Patient with fulminate hepatic failure
* Re-do OLT
* Simultaneous other organ transplant (i.e., pancreas, heart, and small bowel)
* Pre-existing renal failure requiring hemodialysis or continuous hemofiltration and patient refusal to participate in the study.
* Although, it is extremely uncommon for a patient with hepatic failure to become pregnant due to the pathological effect of hepatic failure on the reproductive system, the policy of Liver Transplantation Service at UPMC is to advise young female not to become pregnant while waiting for OLT. In addition the majority of the patients on the liver transplant waiting list at this institution are above 50 years of age. However, when a female patient of child-bearing potential is called in for OLT and there is a suspicion that she might be pregnant, a blood pregnancy test will be performed as a part of the standard of care for these patients.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2004-07; Primary Completion 2007-04 (Actual); Study Completion 2008-01 (Actual)

PRIMARY OUTCOMES:
improve patient and graft outcome. reduce the incidence of postoperative renal dysfunction | one year

CONTACTS AND LOCATIONS:
Overall Officials: Ibtesam A Hilmi, MB CHB, FRCA, Principal Investigator — University of Pittsburgh Medical Center
Locations (1):
- Unversity of Pittsburgh Medical Center, Pittsburgh, Pennsylvania, United States